CLINICAL TRIAL: NCT06150079
Title: Effect of Individualized PEEP Titration on Postoperative Pulmonary Complications in Elderly Patients Undergoing Major Laparoscopic Surgery- A Multicenter Randomized Controlled Clinical Trial
Brief Title: Individualized PEEP Titration on Postoperative Pulmonary Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai Geriatric Medical Center (Other); Zhongshan Hospital (Xiamen), Fudan University (Other); Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B2023-334R
Record Dates: First submitted 2023-11-11; First posted 2023-11-29 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pulmonary Complications; Positive End-expiratory Pressure; Elderly; Laparoscopic Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): After endotracheal intubation, an esophageal balloon is placed and calibrated for accurate positioning and inflation pressure. Continuous monitoring of end-expiratory esophageal pressure (Pes) is conducted. Fixed PEEP of 3 cmH2O is applied throughout the procedure without lung recruitment maneuvers.
- Pes-Guided Group (Experimental): After endotracheal intubation, an esophageal balloon is placed and calibrated for accurate positioning and inflation pressure. Continuous monitoring of end-expiratory esophageal pressure (Pes) is conducted. Lung recruitment is performed at each time point. After lung recruitment, ventilation is adjusted based on the target PEEP. PEEP is chosen to maintain a positive transpulmonary pressure at end-expiration (PL = PEEP - Pes). PEEP titration following lung recruitment should be performed within 1 hour after endotracheal intubation or any procedure that may cause lung collapse, such as pneumoperitoneum, deflation or inflation of the endotracheal tube cuff, changes in position, or endotracheal suctioning.
  Interventions: Procedure: Pes-Guided PEEP titration

INTERVENTIONS:
Procedure: Pes-Guided PEEP titration — Lung recruitment is performed at each time point, involving a switch from volume-controlled (VCV) mode to pressure-controlled (PCV) mode with a pressure setting of 20 cmH2O, RR of 15 bpm, I:E ratio of 1:1, FiO2 of 0.4, and PEEP of 5 cmH2O. During lung recruitment, PEEP is gradually increased in increments of 5 cmH2O, maintained for 5 respiratory cycles until PEEP reaches 20 cmH2O and airway pressure reaches 40 cmH2O, and then maintained for 10 respiratory cycles. After lung recruitment, ventilation is adjusted based on the target PEEP. Each PEEP titration should ensure adequate muscle relaxation, volume status, and hemodynamic stability. PEEP is chosen to maintain a positive transpulmonary pressure at end-expiration (PL = PEEP - Pes). Each PEEP titration should ensure adequate muscle relaxation, volume status, and hemodynamic stability.
  Arms: Pes-Guided Group

SUMMARY:
This study aims to investigate the effectiveness and safety of implementing a personalized positive end-expiratory pressure (PEEP) management strategy guided by esophageal pressure (Pes), as well as its potential to reduce the occurrence of postoperative pulmonary complications (PPCs) in elderly patients undergoing laparoscopic surgery.

DETAILED DESCRIPTION:
This trial is a single-blind, randomized, controlled, multicenter study. Elderly patients undergoing laparoscopic surgery under general anesthesia will be recruited according the inclusion and exclusion criteria. Participants in this study will be randomly assigned into two groups. The total sample size will be 232, with 116 participants in the experimental group and 116 participants in the control group. A stratified block randomization method will be employed, using the ARISCAT score for PPCs risk assessment and individual study centers as stratification factors. Anesthesia routine will be applied during pre-anesthetic preparation, anesthetic induction, maintenance and emergence except intraoperative respiratory management. In the control group, fixed PEEP of 3 cmH2O is applied throughout the procedure without lung recruitment maneuvers. While in the experimental group (Pes-Guided Group), continuous monitoring of end-expiratory esophageal pressure (Pes) is conducted. PEEP is chosen to maintain a positive transpulmonary pressure at end-expiration (PL = PEEP - Pes) after lung recruitment. PEEP titration following lung recruitment should be performed after endotracheal intubation or any procedure that may cause lung collapse, such as pneumoperitoneum, deflation or inflation of the endotracheal tube cuff, changes in position, or endotracheal suctioning. PEEP Titration is also required every hour after the establishment of pneumoperitoneum. Patients will be followed up within 7 days after surgery to assess basic vital signs, potential postoperative pulmonary complications (PPCs). Additionally, postoperative non-respiratory complications will be evaluated. Laboratory tests, the 15-item Quality of Recovery-15 (QoR-15) questionnaire, complications within 30 days after surgery, and 90-day survival rates will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 65 years or older, male or female
2. Scheduled to perform major laparoscopic surgery under general anesthesia
3. Expected duration of surgery ≥ 2 hours
4. Written informed consent is obtainable either from the patient or from a legal surrogate

Exclusion Criteria:

1. BMI ≥ 35 kg/m2.
2. History of pulmonary surgery (of any type).
3. History of severe chronic obstructive pulmonary disease (COPD) requiring non-invasive ventilation and/or home oxygen therapy.
4. Patients on systemic corticosteroid treatment for acute chronic obstructive pulmonary disease exacerbation.
5. Severe pulmonary arterial hypertension, defined as systolic pulmonary artery pressure > 40 mmHg.
6. Heart failure according to the New York Heart Association classification (class III or IV), ongoing hemodynamic instability, or severe shock (determined by the attending internist, cardiac index < 2.5 L/min/m2, or the requirement for positive inotropic drugs to maintain blood pressure).
7. Severe cardiac disease (acute coronary syndrome according to Canadian Cardiovascular Society, atrial flutter/fibrillation, sustained ventricular tachyarrhythmias, metabolic equivalent of tasks (METs) < 4) (METs < 4, determined by the inability to climb ≥ 2 flights of stairs).
8. Severe liver or renal dysfunction (Child-Pugh score 10-15, serum creatinine ≥ 2 mg/dL, or patients requiring peritoneal dialysis or hemodialysis).
9. Neuromuscular disease (of any type).
10. History of bone marrow transplantation or recent history of immunosuppressive drugs (chemotherapy or radiotherapy within 2 months before surgery).
11. Mechanical ventilation duration > 30 minutes within the past 30 days (e.g., surgery under general anesthesia).
12. Requirement for one-lung ventilation.
13. History of acute respiratory distress syndrome with potential need for prolonged postoperative mechanical ventilation.
14. Planned re-intubation after surgery.
15. Pregnancy (excluded by medical history and/or laboratory tests).
16. Brain injury or tumor.
17. Requirement for prone or lateral position during surgery.
18. Severe esophagogastric varices.
19. Enrollment in other interventional studies or refusal to sign informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2025-02-09 (Actual)

PRIMARY OUTCOMES:
postoperative pulmonary complications | within 7 days after surgery
  the incidence of postoperative pulmonary complications

SECONDARY OUTCOMES:
airway peak pressure (cmH2O) | intraoperative
  intraoperative mechanical ventilation parameters
plateau pressure | intraoperative
  intraoperative mechanical ventilation parameters
positive end-expiratory pressure | intraoperative
  intraoperative mechanical ventilation parameters
esophageal pressure (Pes) | intraoperative
  a classical and most widely used marker of pleural pressure which is usually measured by air-filled balloons
driving pressure (cmH2O) | intraoperative
  intraoperative mechanical ventilation parameters
transpulmonary pressure (PL) | intraoperative
  equal to the difference between alveolar pressure and pleural pressure
dynamic lung compliance (mL/cmH20) | intraoperative
  Cdyn = Vt/(Ppeak - PEEP)
static compliance (mL/cmH20) | intraoperative
  pulmonary compliance measured at a fixed volume with no airflow and fully relaxed muscles. static compliance = VT / (Pplat - PEEP)
PaO2/FiO2 ratio | before surgery, intraoperative, and in post-anesthetic care unit
  the ratio of partial pressure of oxygen in arterial blood (PaO2) to the fraction of inspiratory oxygen concentration (FiO2), measured through blood gas analysis
non-respiratory complications | within 7 days after surgery
  the incidence of stroke, myocardial infarction, acute renal failure, DIC, SIRS, sepsis, septic shock, wound infection
QoR-15 scores | day 1 and day 7 after surgery, the day of discharge
  early quality of recovery
unplanned reintubation | day 1 to day 7 after surgery
  the incidence of unplanned reintubation
unplanned transfer to the ICU | day 1 to day 7 after surgery
  the incidence of unplanned transfer to the ICU
duration of ICU stay | day 1 after surgery to the day of discharge, assessed up to 90 days
  duration of ICU stay
length of hospital stay | from the day of admission to the day of discharge, assessed up to 90 days
  the number of days from a patient's hospital admission to discharge
Interleukin-6 level | before surgery, before the end of surgery and in post-anesthetic care unit
  biological indices, result from blood sample
Clara cell secretory protein-16 level | before surgery, before the end of surgery and in post-anesthetic care unit
  biological indices, result from blood samples
soluble receptor for advanced glycation end product level | before surgery, before the end of surgery and in post-anesthetic care unit
  biological indices, result from blood samples
angiopoietin-2 level | before surgery, before the end of surgery and in post-anesthetic care unit
  biological indices, result from blood samples
plasminogen activator inhibitor-1 | before surgery, before the end of surgery and in post-anesthetic care unit
  biological indices, result from blood samples
mortality rates | at 90 days after surgery
  mortality rates
complications | at 30 days after surgery
  including postoperative respiratory and non-respiratory complications
vital signs | admission to operating room to day 7 after surgery, and the day of discharge
  vital signs will be recorded at any key time points from admission to operating room to extubation
Vasoactive medications dosages | intraoperative
  Vasoactive medications includes norepinephrine, phenylephrine, ephedrine

CONTACTS AND LOCATIONS:
Overall Officials: Changhong Miao, Study Director — Zhongshang Hospital Fudan University; Jing Zhong, Principal Investigator — Zhongshang Hospital Fudan University
Locations (4):
- China (4):
  - 180 Fenglin Road, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Geriatric Medical Center, Shanghai
  - Zhongshan Hospital (Xiamen), Fudan University, Xiamen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data generated during the study will be made available on reasonable request to qualified researchers, following publication of the primary results, and in accordance with institutional and ethical guidelines.

REFERENCES:
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Hegeman MA, Hemmes SN, Kuipers MT, Bos LD, Jongsma G, Roelofs JJ, van der Sluijs KF, Juffermans NP, Vroom MB, Schultz MJ. The extent of ventilator-induced lung injury in mice partly depends on duration of mechanical ventilation. Crit Care Res Pract. 2013;2013:435236. doi: 10.1155/2013/435236. Epub 2013 Apr 17. PMID 23691294
- [Background] Tusman G, Bohm SH, Warner DO, Sprung J. Atelectasis and perioperative pulmonary complications in high-risk patients. Curr Opin Anaesthesiol. 2012 Feb;25(1):1-10. doi: 10.1097/ACO.0b013e32834dd1eb. PMID 22113182
- [Background] Fernandez-Bustamante A, Frendl G, Sprung J, Kor DJ, Subramaniam B, Martinez Ruiz R, Lee JW, Henderson WG, Moss A, Mehdiratta N, Colwell MM, Bartels K, Kolodzie K, Giquel J, Vidal Melo MF. Postoperative Pulmonary Complications, Early Mortality, and Hospital Stay Following Noncardiothoracic Surgery: A Multicenter Study by the Perioperative Research Network Investigators. JAMA Surg. 2017 Feb 1;152(2):157-166. doi: 10.1001/jamasurg.2016.4065. PMID 27829093
- [Background] Ferrando C, Soro M, Unzueta C, Suarez-Sipmann F, Canet J, Librero J, Pozo N, Peiro S, Llombart A, Leon I, India I, Aldecoa C, Diaz-Cambronero O, Pestana D, Redondo FJ, Garutti I, Balust J, Garcia JI, Ibanez M, Granell M, Rodriguez A, Gallego L, de la Matta M, Gonzalez R, Brunelli A, Garcia J, Rovira L, Barrios F, Torres V, Hernandez S, Gracia E, Gine M, Garcia M, Garcia N, Miguel L, Sanchez S, Pineiro P, Pujol R, Garcia-Del-Valle S, Valdivia J, Hernandez MJ, Padron O, Colas A, Puig J, Azparren G, Tusman G, Villar J, Belda J; Individualized PeRioperative Open-lung VEntilation (iPROVE) Network. Individualised perioperative open-lung approach versus standard protective ventilation in abdominal surgery (iPROVE): a randomised controlled trial. Lancet Respir Med. 2018 Mar;6(3):193-203. doi: 10.1016/S2213-2600(18)30024-9. Epub 2018 Jan 19. PMID 29371130
- [Background] Zhang C, Xu F, Li W, Tong X, Xia R, Wang W, Du J, Shi X. Driving Pressure-Guided Individualized Positive End-Expiratory Pressure in Abdominal Surgery: A Randomized Controlled Trial. Anesth Analg. 2021 Nov 1;133(5):1197-1205. doi: 10.1213/ANE.0000000000005575. PMID 34125080
- [Background] Akoumianaki E, Maggiore SM, Valenza F, Bellani G, Jubran A, Loring SH, Pelosi P, Talmor D, Grasso S, Chiumello D, Guerin C, Patroniti N, Ranieri VM, Gattinoni L, Nava S, Terragni PP, Pesenti A, Tobin M, Mancebo J, Brochard L; PLUG Working Group (Acute Respiratory Failure Section of the European Society of Intensive Care Medicine). The application of esophageal pressure measurement in patients with respiratory failure. Am J Respir Crit Care Med. 2014 Mar 1;189(5):520-31. doi: 10.1164/rccm.201312-2193CI. PMID 24467647
- [Background] Fernandez-Bustamante A, Sprung J, Parker RA, Bartels K, Weingarten TN, Kosour C, Thompson BT, Vidal Melo MF. Individualized PEEP to optimise respiratory mechanics during abdominal surgery: a pilot randomised controlled trial. Br J Anaesth. 2020 Sep;125(3):383-392. doi: 10.1016/j.bja.2020.06.030. Epub 2020 Jul 16. PMID 32682559
- [Background] Cammarota G, Lauro G, Sguazzotti I, Mariano I, Perucca R, Messina A, Zanoni M, Garofalo E, Bruni A, Della Corte F, Navalesi P, Bignami E, Vaschetto R, Mojoli F. Esophageal Pressure Versus Gas Exchange to Set PEEP During Intraoperative Ventilation. Respir Care. 2020 May;65(5):625-635. doi: 10.4187/respcare.07238. PMID 32345760
- [Derived] Zhong J, Xu P, Zhou X, Zou K, Yu J, Liu Y, Zhu M, Wei M, Yang H, Miao C. Effect of intraoperative oesophageal pressure-guided PEEP on postoperative pulmonary complications in elderly patients undergoing major laparoscopic surgery: study protocol for a multicentre randomised controlled clinical trial in China. BMJ Open. 2025 Aug 13;15(8):e096219. doi: 10.1136/bmjopen-2024-096219. PMID 40812804